CLINICAL TRIAL: NCT05308355
Title: Evaluation of an "Opioid Free Anesthesia" Protocol in Thoracoscopic Carcinological Thoracic Surgery
Brief Title: Opioid-free Anesthesia and Thoracoscopy Surgery
Acronym: OFAT
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC22_0112
Record Dates: First submitted 2022-02-15; First posted 2022-04-04 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Opioid Free Anesthesia; Thoracic Surgery
Keywords: Video-thoracoscopy; Chronic Pain; Opioid Free Anesthesia; Thoracic surgery
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OFA : Opioid Free Anesthesia: Opioid-free surgery. Analgesia provided by attenuation analgesic 1, dexmedetomidine, ketamine and general anesthesia by propofol. Regional loco anesthesia is performed in the OFA group and possible in the OBA group. It's local service protocol used since 1 year.
- OBA : Opioid Based Anesthesia: Conventional anesthesia with Propofol and Sufentanil boli with the possibility of regional loco anesthesia.

SUMMARY:
Evaluation of a service OFA (Opioid-free Anesthesia) protocol on post-operative pain of patients operated on by video-thoracoscopic carcinologic surgery by counting them to a group of patients receiving standard general anesthesia with opioid.

DETAILED DESCRIPTION:
A service protocol based on opioid-free anesthesia in patients undergoing pulmonary carcinologic surgery under video-thoracoscopy will be evaluated.

The investigative team want to recruit 100 patients prospectively. These patients will be randomly assigned on the day of surgery between OFA (Opioid Free Anesthesia) and OBA (Opioid Based Anesthesia).

Anesthesia and analgesia of patients in the OFA group will be performed without morphine according to the validated local protocol. We will use level 1 and 2 analgesics (paracetamol, NSAIDs and nefopam) associated with an erector spine block and anesthesia under propofol, dexmedetomidine and ketamine ivse.

Patients in the OBA group will have so-called "basic" anesthesia and analgesia with opioids according to usual practice.

Postoperative pain by collecting morphine consumption in the first 48 hours postoperatively between the two groups will be compared.

Chronic neuropathic postoperative pain will also be collected by a telephone questionnaire at 3 months postoperative.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Patient operated on pulmonary carcinologic surgery by thoracoscopy of a foreseeable duration greater than 2 hours

Exclusion Criteria:

* Patient with unstable unstable unstable coronary artery disease,
* Patient contraindicated for the use of dexmedetomidine: heart rate<50 / min, High degree atrioventricular block (2 and 3) unless fitted (carrier of a pacemaker),
* Patient on beta-blocker, allergy to Dexdor®,
* Patient allergic to other drugs used in OFA (Paracetamol and NSAIDs).
* Renal insufficiency patient with creatinine clearance<30ml/min will not be excluded but will not receive NSAIDs.
* Minor patient,
* Adult patient under guardianship or curators.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing lung oncology surgery under video-thoracoscopy lasting more than 2 hours.
  Patients will be randomly assigned to a group without a random draw. Only the anesthesiologist trained at the OFA will be able to do the OFA
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Day 2
  Total morphine consumption over the first 48 post operative hours in milligrammes

SECONDARY OUTCOMES:
Preoperatory haemodynamic tolerance | Day 0
  Maximum doses of norepinephrine intraoperatively in µg/kg/min.
Quality of intraoperative anesthesia | Day 0
  Duration of surgery (time between entering the operating room and leaving the room) in minutes.
Ileus Postoperative | Day 4
  Presence of postoperative ileus (defined by the presence 2 of the following criteria from the 4th postoperative day: nausea and vomiting, absence of food recovery, no stool or gas in the last 24 hours, abdominal meteorism, radiological arguments)
Duration of hospitalization | Day 10
  Length of hospitalization (Time between arrival at the hospital and discharge) in days.
Chronic neuropathic pain | Month-3
  Evaluation of neuropathic pain (assessed by the DN 4 score:diagnosis of neuropathic pain)
Long-term morphine consumption | Month-3
  Morphine consumption at 3-month (yes/no)
Physical form recovery | Month-3
  Time between surgery and resumption of physical activity in days.

CONTACTS AND LOCATIONS:
Overall Officials: Julien CADIET, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No